CLINICAL TRIAL: NCT01663311
Title: Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) With Double-Cone-Coil in Patients With Chronic Tinnitus (Ti-CDC)
Brief Title: Repetitive Transcranial Magnetic Stimulation With Double Cone Coil in Chronic Tinnitus
Acronym: Ti-CDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, Ph.D., University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Uni-Reg-Ti-CDC01
Record Dates: First submitted 2012-07-23; First posted 2012-08-13 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Tinnitus
Keywords: rTMS; repetitive transcranial magnetic stimulation; chronic tinnitus; subjective tinnitus; double cone coil
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medial Frontal rTMS Double-Cone-Coil (Experimental): High frequency rTMS ( Alpine Biomed Mag Pro Option) applied over medial superior frontal cortex (supplementary motor cortex) (Brodman area 6/8),Double-Cone-water-cooled-Coil (2000 Stimuli of 10 Hz each session), 110% motor threshold; followed by: low frequency rTMS ( Alpine Biomed Mag Pro Option) applied over left temporoparietal cortex, Butterfly-water-cooled-Coil (2000 Stimuli of 1 Hz each session), 110% motor threshold.
  Interventions: Device: Medial Frontal rTMS Double-Cone-Coil
- Left DLPFC Butterfly Coil (Experimental): High frequency rTMS ( Alpine Biomed Mag Pro Option): 2000 stimuli of 20 Hz over the left DLPFC (each session), Butterfly-water-cooled-Coil, 110% motor threshold; followed by: low frequency rTMS ( Alpine Biomed Mag Pro Option) applied over left temporoparietal cortex, Butterfly-water-cooled-Coil (2000 Stimuli of 1 Hz each session), 110% motor threshold.
  Interventions: Device: Left DLPFC Butterfly Coil

INTERVENTIONS:
Device: Medial Frontal rTMS Double-Cone-Coil — High frequency rTMS ( Alpine Biomed Mag Pro Option) applied over medial superior frontal cortex (supplementary motor cortex) (Brodman area 6/8),Double-Cone-water-cooled-Coil (2000 Stimuli of 10 Hz each session), 110% motor threshold; followed by: low frequency rTMS ( Alpine Biomed Mag Pro Option) applied over left temporoparietal cortex, Butterfly-water-cooled-Coil (2000 Stimuli of 1 Hz each session), 110% motor threshold.
  Arms: Medial Frontal rTMS Double-Cone-Coil
Device: Left DLPFC Butterfly Coil — High frequency rTMS ( Alpine Biomed Mag Pro Option): 2000 stimuli of 20 Hz over the left DLPFC (each session), Butterfly-water-cooled-Coil, 110% motor threshold; followed by: low frequency rTMS ( Alpine Biomed Mag Pro Option) applied over left temporoparietal cortex, Butterfly-water-cooled-Coil (2000 Stimuli of 1 Hz each session), 110% motor threshold.
  Arms: Left DLPFC Butterfly Coil

SUMMARY:
Transcranial Magnetic Stimulation is used to modulate both the auditory neural pathways contributing to the perception of phantom sounds, and the regulatory neural network responsible for the generation of the individual amount of suffering caused by chronic tinnitus.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. Treatment remains difficult. Most available therapies focus on habituation rather than treating the cause. Tinnitus has been shown to be generated in the brain, as a result of functional reorganization of auditory neural pathways and tonotopic maps in the central auditory system. Low-frequency rTMS applied to the temporoparietal areas has been investigated for the treatment of hyperexcitability disorders such as auditory hallucinations and tinnitus. Pilot data indicate that taking into account affective components of the multiple overlapping neural networks responsible for the generation of a bothersome subjective tinnitus might enhance the efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) treatment in chronic tinnitus. A newly developed coil, the so-called double cone coil will be examined with regard to feasibility, safety and clinical efficacy in patients suffering from chronic tinnitus in a controlled pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bothersome, subjective chronic tinnitus
* Duration of tinnitus more than 6 months

Exclusion Criteria:

* Objective tinnitus
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery;
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Prior treatment with TMS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of treatment responders (TQ reduction > 5, contrast Baseline versus end of treatment/ day 12) | Day 12

SECONDARY OUTCOMES:
Change of tinnitus severity as measured by the Tinnitus Questionaire of Goebel&Hiller, Tinnitus Handicap Inventory (THI), Tinnitus Severity Scale and TBF-12 | Baseline vs. day 90
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Baseline vs. day 90
Change in quality of life as measured by the WHOQoL | Baseline vs. day 90

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Ph.D., Principal Investigator — University of Regensburg, Dept of Psychiatry
Locations (1):
- University of Regensburg- Dept of Psychiatry, Regensburg, Germany